CLINICAL TRIAL: NCT00901888
Title: Investigating the Interaction of Apelin and Angiotensin II Peripheral Resistance Vessels in Vivo in Man
Brief Title: Interaction of Apelin and Angiotensin in the Human Forearm Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Dr Gareth Barnes, Research Fellow, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FS/09/019/26905 - 1a
Record Dates: First submitted 2009-05-08; First posted 2009-05-14 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Heart Disease; Vasodilation
Keywords: Renin Angiotensin System
MeSH Terms: conditions — Heart Diseases; Aneurysm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angiotensin II infusion (Experimental): Using forearm venous occlusion plethysmography angiotensin II will be infused to cause reduction in forearm blood flow. Infusion of apelin and sodium nitroprusside will given and vasodilatation will be assessed. Blood samples for the infused arm and contra-lateral arm will be taken at regular time points to assess local and systemic changes in relevant hormones.
  Interventions: Drug: Apelin infusion; Drug: Sodium nitroprusside infusion
- Noradrenaline (Active Comparator): Using forearm venous occlusion plethysmography noradrenaline will be infused to cause reduction in forearm blood flow. Infusion of apelin and sodium nitroprusside will given and vasodilatation will be assessed. Blood samples for the infused arm and contra-lateral arm will be taken at regular time points to assess local and systemic changes in relevant hormones.
  Interventions: Drug: Apelin infusion; Drug: Sodium nitroprusside infusion

INTERVENTIONS:
Drug: Apelin infusion — Infusion of up to 10picmol/min will be administered intra-arterially to induce vasoconstriction. Thereafter infusions of apelin (0.1, 1.0, 3.0nmol/min) will be given for 6mins each. During the same study, sodium nitroprusside will given (1.0, 2.0, 4.0 microg/min) for 6mins.
Drug: Sodium nitroprusside infusion — Infusion of up to 150-600picmol/min will be administered intra-arterially to induce vasoconstriction. Thereafter infusions of apelin (0.1, 1.0, 3.0nmol/min) will be given for 6mins each. During the same study, sodium nitroprusside will given (1.0, 2.0, 4.0 microg/min) for 6mins.

SUMMARY:
The apelin-APJ system is a relatively new discovery. It has generated interest in part due to it's apparent ability to counteract the renin-angiotensin system, which is frequently overactive in many cardiovascular disease.

Angiotensin has a powerful ability to cause blood vessels constrict and reduces their diameter. One of the actions of apelin is to cause blood vessels to relax and the investigators specifically wish test the hypothesis that apelin will cause blood vessels constricted by angiotensin II to relax.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old

Exclusion Criteria:

* Lack of informed consent
* Age < 18 years,
* Current involvement in other research studies,
* Systolic blood pressure >190 mmHg or <100 mmHg
* Malignant arrhythmias
* Renal or hepatic failure
* Haemodynamically significant aortic stenosis
* Severe or significant co morbidity
* Women of childbearing potential.
* Any regular medication
* Previous history of any cardiovascular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in apelin mediated forearm blood flow | 12 months

SECONDARY OUTCOMES:
Change in local and systemic plasma apelin concentration in response angiotensin II infusion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gareth D Barnes, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Clincial Research Facility, Royal Infirmary of Edinburgh, 51 Little France Cresc, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Barnes GD, Alam S, Carter G, Pedersen CM, Lee KM, Hubbard TJ, Veitch S, Jeong H, White A, Cruden NL, Huson L, Japp AG, Newby DE. Sustained cardiovascular actions of APJ agonism during renin-angiotensin system activation and in patients with heart failure. Circ Heart Fail. 2013 May;6(3):482-91. doi: 10.1161/CIRCHEARTFAILURE.111.000077. Epub 2013 Mar 21. PMID 23519586